CLINICAL TRIAL: NCT00880399
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Fixed Dose Study Evaluating the Efficacy and Safety of Orvepitant in Subjects With Major Depressive Disorder
Acronym: orvepitant MDD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: To allow assessment of isolated events of seizure during program
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 111733
Record Dates: First submitted 2009-04-09; First posted 2009-04-13 (Estimated); Results first posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-04

CONDITIONS: Depressive Disorder, Major
Keywords: depression; QIDS-SR; HAMD-17; orvepitant; MDD; neurokinin-1 antagonist; double-blind; Phase II; randomized; efficacy; placebo; safety
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — orvepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): inactive placebo to match orvepitant 30 and 60 mg dosage forms
  Interventions: Other: placebo
- Orvepitant 30 mg (Experimental): 30 mg/day (low dose)
  Interventions: Drug: orvepitant
- Orvepitant 60 mg (Experimental): 60 mg/day (high dose)
  Interventions: Drug: orvepitant

INTERVENTIONS:
Drug: orvepitant — Neurokinin-1 (NK-1) antagonist
  Other Names: GW823296
  Arms: Orvepitant 30 mg; Orvepitant 60 mg
Other: placebo — inactive placebo to match orvepitant 30 and 60 mg dosage forms
  Arms: Placebo

SUMMARY:
This is a 6-week, randomised, multicenter, double-blind, placebo controlled, fixed dose parallel group study to assess the efficacy and safety of orvepitant (30 and 60 mg/day) versus placebo in subjects with a diagnosis of a Major Depressive Disorder, whose symptoms are considered moderate or severe.

Following an initial screening visit, subjects fulfilling the study inclusion and exclusion criteria will enter a pre-treatment screening phase to permit evaluation of the laboratory and ECG assessments and to confirm eligibility for inclusion into the study. This screening phase will be a minimum of 7 days, but no longer than 21 days. At the completion of the screening period, eligible subjects will be randomised at the baseline visit to receive either orvepitant 30mg/day, orvepitant 60mg/day or placebo (equal chance of receiving any of the three possible treatments, i.e., a 1:1:1 ratio) for a six-week double-blind treatment phase. Those subjects randomised to receive placebo will receive study medication identical in appearance to that received by subjects assigned to receive orvepitant 30 or 60mg/day.

Efficacy will be assessed via standard depression symptom and severity rating scales or questionaires. The Hamilton Depression Rating Scale (HAM-D) will be used as the primary measure. Secondary efficacy endpoints include the Quick Inventory of Depressive Symptomatology (QIDS-SR) and the Clinical Global Impression- Global Improvement and Severity of Illness Scale (CGI-I and CGI-S, respectively).

Safety will be assessed by monitoring for adverse events (side effects) and through periodic laboratory evaluations (blood tests), vital signs assessments (e.g., blood pressure, heart rate, temperature) and heart function measurements (electrocardiograms, or ECGs).

DETAILED DESCRIPTION:
The purpose of the current study is to test the safety and the anti-depressant effects of orvepitant, an investigational antidepressant. Efficacy will be assessed using standard depression symptom and severity rating scales (questionaires). The Hamilton Depression Rating Scale (HAM-D) will serve as the primary measure of efficacy, and . Secondary efficacy endpoints include the Bech Melancholia Scale (sum of items 1, 2, 7, 8, 10, and 13 of the 17-item HAM-D scale), the Quick Inventory of Depressive Symptomatology (QIDS-SR), the Clinical Global Impression- Global Improvement and Severity of Illness Scale (CGI-I and CGI-S, respectively), the HAM-D anxiety factor score (sum of items 10, 11, 12, 13, 15 and 17), the Cognitive and Physical Function Questionnaire (CPFQ) and a morning sleep questionnaire.

Safety and tolerability will be assessed by monitoring adverse events (AEs or side effects), physical examinations (including vital signs such as blood pressure and heart rate), clinical laboratory assessments (blood tests), electrical recordings of the heart (electrocardiograms or ECG's), the Columbia Suicidality Severity Rating Scale (CSSRS), Sexual Function Questionnaire (SFQ), and weight change.

Blood samples will be taken at different time points to assess blood levels of orvepitant in patients, allowing the relationship between amount of orvepitant in the body and efficacy to be studied.

The primary objective of the study is to evaluate the antidepressant efficacy of orvepitant (30 and 60mg/day) versus placebo (a "sugar pill", with no active ingredients). The secondary objectives include assessing the safety and tolerability of orvepitant, assessing the profile of appearance and disappearance of orvepitant in the body (blood) following administration (i.e., assessing how long the drug remains in the body), and lastly to examine the relationship between blood levels of the drug and efficacy (i..e, the change in HAM-D total score relative to what it was before starting the study medication.

Following an initial screening visit, subjects fulfilling the study entrance criteria will enter a pre-treatment screening phase to permit evaluation of the laboratory and electrocardiogram assessments and to confirm eligibility for inclusion into the study. This screening phase will be a minimum of 7 days, but no longer than 21 days. During the screening period, subjects may undergo up to three different assessments of their depressive symptoms, this may occur via a face-to-face interview or via an interview over the telephone. Upon completion of the screening period, eligible subjects will be randomly assigned at the baseline visit to one of three treatment regimens: orvepitant 30mg/day, orvepitant 60mg/day or placebo for a six-week treatment phase. The chances of receiving each of the three possible treatments will be equal. Orvepitant will be administered as tablets. Those subjects randomised to receive placebo will receive study medication identical in appearance to that received by subjects assigned to receive orvepitant.

During the treatment phase, subjects will be required to return to the clinic at the end of Weeks 1, 2, 4 and 6. In addition, all subjects will be required to return for a follow-up visit 14 days after the last dose of study medication. In addition, all subjects with ongoing adverse events at the 14-day follow-up visit will be required to return for a further follow-up visit 28 days after the last dose of study medication.

Male and female outpatients between the ages of 18 to 64 years inclusive with a primary diagnosis of Major Depressive Disorder will be enrolled into this study. A total of approximately 350 subjects are expected to be enrolled at approximately 20 different study sites in the U.S. and Canada.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have the ability to comprehend the Informed Consent Form.
* Male or female outpatients, aged 18-64, inclusive.
* A primary diagnosis of major depressive disorder, single episode or recurrent
* Subjects must, in the investigator's opinion and based on the subject's history, have met depression criteria for at least 8 weeks prior to the Screening Visit.
* Subjects with symptom severity considered to be at least moderate to severe by the investigator.
* Women of childbearing potential are only eligible IF they commit to consistent and correct use of an acceptable method of birth control that must be documentation at each visit

Exclusion Criteria:

* Subjects whose mood-related symptoms are better accounted for by a diagnosis other than depression; subjects diagnosed with Alzheimer's Disease or other form of dementia; subjects diagnosed with a current/recent eating disorder such as anorexia nervosa or bulimia; subjects with a diagnosed history of schizophrenia, schizoaffective disorder, or Bipolar Disorder.
* Subjects with any history of a significant abnormality of the neurological system (including dementia and other cognitive disorders or significant head injury) or any history of seizures (convulsions).
* Subjects have a positive urine test at screening for illegal drug use and/or who have a history of substance abuse or dependence (alcohol or drugs) within the past 12 months.
* Subjects who are currently receiving regularly scheduled psychotherapy (individual or group), plan to start psychotherapy during the trial or have received regularly scheduled psychotherapy during the 12 week period prior to the Screening Visit.
* Subjects who have a history of failing to respond to adequate treatment with an antidepressant, i..e, failure to improve following administration of at least two other antidepressants, each given for at least 4 weeks.
* Subjects who, in the investigator's judgement, pose a homicidal or serious suicidal risk, have made a suicide attempt within the 6 months preceding screening or who have ever been homicidal.
* Subjects who have received the following treatments for depression in the past: electroconvulsive therapy (ECT), vagal stimulation, or transcranial magnetic stimulation (TMS) within the 6 months prior to the Screening Visit.
* Subjects with an unstable medical disorder; or with a disorder that otherwise would likely interfere with the activity of the study medication (orvepitant).
* Subjects have any screening laboratory abnormality that in the investigator's judgement is considered to be clinically significant.
* Subjects with an abnormal thyroid test at the Screening Visit. Subjects maintained on thyroid medication must have normal thyroid levels for a period of at least six months prior to the Screening Visit.
* Subjects have any screening electrocardiography (ECG) finding that in the investigator's judgement is considered to be clinically significant.
* Women who have a positive pregnancy test at the Screening Visit, a positive urine dipstick test at the Baseline (Randomization) Visit, or who are lactating or planning to become pregnant within the 4 months following the Screen Visit.
* Subjects who have taken other psychoactive drugs within two weeks prior to the Baseline Visit i.e. at any time during the Screening period. This includes "over-the-counter" psychoactive medications such as St. John's Wort and SAM-e.
* Subjects who have taken other drugs within 2 weeks prior to the Baseline visit which the investigator feels may interact with the study medication.
* Subjects who are currently participating in another clinical trial in which the subject is or will be exposed to an investigational or non-investigational drug or device, or has done so within the preceding month for studies unrelated to depression, or 6 months for studies related to depression.
* Subjects who have no contact with an adult on a daily basis. This would exclude subjects who are not living with at least one other adult or subjects who do not have an adult who contacts them on a daily basis.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 328 (Actual)
Dates: Start 2009-03-01; Primary Completion 2010-06-01 (Actual); Study Completion 2010-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (20):
- United States (17):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Arcadia, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, National City, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Bradenton, Florida
  - GSK Investigational Site, Maitland, Florida
  - GSK Investigational Site, North Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Lincoln, Rhode Island
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Middleton, Wisconsin
- Canada (3):
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario

REFERENCES:
- [Background] Ratti E, Bettica P, Alexander R, Archer G, Carpenter D, Evoniuk G, Gomeni R, Lawson E, Lopez M, Millns H, Rabiner EA, Trist D, Trower M, Zamuner S, Krishnan R, Fava M. Full central neurokinin-1 receptor blockade is required for efficacy in depression: evidence from orvepitant clinical studies. J Psychopharmacol. 2013 May;27(5):424-34. doi: 10.1177/0269881113480990. Epub 2013 Mar 28. PMID 23539641

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 20 centers across the United States of America (USA) (17 centers) and Canada (3 centers) from 04 March 2009 to 16 June 2010.
Pre-assignment Details: A total of 787 participants were screened for study eligibility, of which 331 participants were randomized. Out of 331 participants, 3 did not receive the study medication. All subjects population included all participants who had received at least one dose of the study medication and comprised of 328 participants.
Groups:
- Placebo: Participants received Orvepitant matching placebo tablets via oral route, once daily in the evening, for a total of 6 weeks.
- Orvepitant 30 mg: Participants received Orvepitant 30 mg tablets via oral route, once daily in the evening, for a total of 6 weeks.
- Orvepitant 60 mg: Participants received Orvepitant 60 mg tablets via oral route, once daily in the evening, for a total of 6 weeks.
Period: Overall Study
Arm/Group | Placebo | Orvepitant 30 mg | Orvepitant 60 mg
Started | 108 | 113 | 107
Completed | 77 | 84 | 81
Not Completed | 31 | 29 | 26
Not completed — Adverse Event | 4 | 6 | 5
Not completed — Lack of Efficacy | 1 | 4 | 2
Not completed — Protocol Violation | 4 | 4 | 6
Not completed — Study closed/terminated | 3 | 7 | 4
Not completed — Lost to Follow-up | 8 | 5 | 3
Not completed — Physician Decision | 5 | 0 | 3
Not completed — Withdrawal by Subject | 6 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Orvepitant 30 mg | Orvepitant 60 mg | Total
Number analyzed (Participants) | 108 | 113 | 107 | 328
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.7 (11.67) | 41.0 (11.45) | 38.2 (11.15) | 39.7 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 68 | 70 | 214
  Male | 32 | 45 | 37 | 114
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2 | 4
  Asian | 4 | 2 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 16 | 17 | 21 | 54
  White | 86 | 92 | 79 | 257
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the 17-item Hamilton Depression Rating Scale (HAM-D) Total Score
Description: The HAM-D is designed to measure severity of depressive symptoms in participants with primary depressive illness. The scale is a checklist of items (1: depressed mood, 2: feelings of guilt, 3: suicide, insomnia early, 4: insomnia early, 5: insomnia middle, 6: insomnia late, 7: work and activities, 8: retardation, 9: agitation, 10: anxiety psychic item 10: anxiety psychic, item 11: anxiety somatic, item 12: somatic symptoms gastrointestinal, 13: somatic symptoms general, 14: genital symptoms, 15: hypochondriasis, 16: loss of weight and 17: insight) that are ranked on a scale of 0 to 4 or 0 to 2 (4 and 2: highly severe and 0: not present). The HAM-D total score is calculated by summing individual response scores on the HAM-D questionnaire. The highest possible score is 52, representing most severe measure of depression; lowest possible score is 0, representing no depression. Baseline was Day 1. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Day 1) to Week 6
Population: The Intent-to-Treat (ITT) population comprised of all participants who were randomized and received at least one dose of double blind medication and for whom at least one post-randomization assessment was available. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | Orvepitant 30 mg | Orvepitant 60 mg
Number analyzed (Participants) | 103 | 110 | 107
Scores on a Scale
  Week 1: number analyzed (Participants) | 102 | 110 | 103
  Week 1 | -3.72 (0.438) | -4.19 (0.417) | -4.87 (0.433)
  Week 2: number analyzed (Participants) | 94 | 102 | 100
  Week 2 | -5.32 (0.540) | -7.21 (0.515) | -7.16 (0.525)
  Week 4: number analyzed (Participants) | 85 | 97 | 93
  Week 4 | -7.40 (0.665) | -9.61 (0.627) | -10.45 (0.641)
  Week 6: number analyzed (Participants) | 78 | 86 | 84
  Week 6 | -9.08 (0.777) | -11.49 (0.735) | -11.93 (0.749)
Statistical Analysis 1: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitatnt 30 mg at Week 1; Test type: Superiority or Other; p = 0.4295, Mixed Models Repeated Measures; Mean Difference (Net) = -0.47, 95% CI 2-sided [-1.65 to 0.70]
Statistical Analysis 2: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitatnt 60 mg at Week 1; Test type: Superiority or Other; p = 0.0586, Mixed Models Repeated Measures; Mean Difference (Net) = -1.15, 95% CI 2-sided [-2.34 to 0.04]
Statistical Analysis 3: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitatnt 30 mg at Week 2; Test type: Superiority or Other; p = 0.0111, Mixed Models Repeated Measures; Mean Difference (Net) = -1.89, 95% CI 2-sided [-3.34 to -0.43]
Statistical Analysis 4: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitatnt 60 mg at Week 2; Test type: Superiority or Other; p = 0.0141, Mixed Models Repeated Measures; Mean Difference (Net) = -1.84, 95% CI 2-sided [-3.30 to -0.37]
Statistical Analysis 5: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitatnt 30 mg at Week 4; Test type: Superiority or Other; p = 0.0152, Mixed Models Repeated Measures; Mean Difference (Net) = -2.22, 95% CI 2-sided [-4.00 to -0.43]
Statistical Analysis 6: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitatnt 60 mg at Week 4; Test type: Superiority or Other; p = 0.0010, Mixed Models Repeated Measures; Mean Difference (Net) = -3.06, 95% CI 2-sided [-4.86 to -1.25]
Statistical Analysis 7: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitatnt 30 mg at Week 6; Test type: Superiority or Other; p = 0.0245, Mixed Models Repeated Measures; Mean Difference (Net) = -2.41, 95% CI 2-sided [-4.50 to -0.31]
Statistical Analysis 8: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitatnt 60 mg at Week 6; Test type: Superiority or Other; p = 0.0082, Mixed Models Repeated Measures; Mean Difference (Net) = -2.86, 95% CI 2-sided [-4.97 to -0.75]

2. Secondary Outcome: Percentage of Participants With a >= 50 Percent (%) Reduction From Baseline in HAM-D Total Score
Description: Participants who had 50% or greater reduction from Baseline in their total HAMD score were termed as responders. The HAM-D was designed to measure the severity of depressive symptoms in participants with primary depressive illness. The scale is a checklist of items that are ranked on a scale of 0 to 4 or 0 to 2. Items with quantifiable severity are scored 0 to 4 (4 indicating the greatest severity) or 0 to 2 (2 indicating the greatest severity) with 0 indicating not present. The HAM-D Total Score is calculated by summing the individual response scores on the HAM-D questionnaire. The highest possible score is 52, which represents the most severe measure of depression; the lowest possible score is 0, which represents an absence of depression. The HAM-D is also useful for monitoring changes in depressive symptoms with treatment and in comparing the efficacy of various interventions if the participant requires more than one type of treatment. Baseline was Day 1.
Time Frame: Baseline (Day 1) to Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Orvepitant 30 mg | Orvepitant 60 mg
Number analyzed (Participants) | 103 | 110 | 107
Percentage of participants
  Week 1: number analyzed (Participants) | 102 | 110 | 103
  Week 1 | 5 | 5 | 4
  Week 2: number analyzed (Participants) | 94 | 102 | 100
  Week 2 | 10 | 15 | 12
  Week 4: number analyzed (Participants) | 85 | 97 | 93
  Week 4 | 19 | 27 | 33
  Week 6: number analyzed (Participants) | 78 | 86 | 84
  Week 6 | 29 | 42 | 39

3. Secondary Outcome: Number of Participants With (Maintained) Clinical Response
Description: Clinical response or antidepressant response was defined as >= 50% reduction from randomization in their HAMD total score, where this response was maintained until the end of the Treatment Phase (Week 6). Participants who met the >= 50% reduction at Week 6 without also having met it at Week 4 were not considered to have reached a maintained response, and therefore were censored at Week 6. Number of participants with maintained clinical response are reported.
Time Frame: Up to Week 6
Population: ITT Population.
Measure: Number; unit: Participants
Arm/Group | Placebo | Orvepitant 30 mg | Orvepitant 60 mg
Number analyzed (Participants) | 103 | 110 | 107
Participants | 13 | 21 | 22
Statistical Analysis 1: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 6; Test type: Superiority or Other; p = 0.51, Log Rank; Hazard Ratio (HR) = 1.60, 95% CI 2-sided [0.80 to 3.19]
Statistical Analysis 2: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 6; Test type: Superiority or Other; p = 0.37, Log Rank; Hazard Ratio (HR) = 1.66, 95% CI 2-sided [0.84 to 3.30]

4. Secondary Outcome: Change From Baseline in the Bech Melancholia Scale Total Score (Sum of Items 1, 2, 7, 8, 10, and 13 of the 17-item HAMD Scale)
Description: The Bech Melancholia is sum of scores on 6 items/questions (item 1: depressed mood, item 2: feelings of guilt, item 7: work and activities, item 8: retardation, item 10: anxiety psychic and item 13: somatic symptoms general) pertaining to melancholia within HAM-D. The items are rated on a scale of 0 to 4 (items 1, 2, 7, 8 and 10) or 0 to 2 (item 13), higher scores reflecting greater severity. The highest possible score is 24, which represents the most severe measure of melancholy; the lowest possible score is 0, which represents an absence of melancholy. Baseline was Day 1. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Day 1) to Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | Orvepitant 30 mg | Orvepitant 60 mg
Number analyzed (Participants) | 103 | 110 | 107
Scores on a Scale
  Week 1: number analyzed (Participants) | 102 | 110 | 103
  Week 1 | -1.68 (0.237) | -1.77 (0.225) | -1.83 (0.233)
  Week 2: number analyzed (Participants) | 94 | 102 | 100
  Week 2 | -2.35 (0.289) | -3.39 (0.276) | -3.26 (0.281)
  Week 4: number analyzed (Participants) | 85 | 97 | 93
  Week 4 | -3.20 (0.366) | -4.49 (0.345) | -4.88 (0.352)
  Week 6: number analyzed (Participants) | 78 | 86 | 84
  Week 6 | -4.30 (0.424) | -5.53 (0.402) | -5.84 (0.409)
Statistical Analysis 1: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 1; Test type: Superiority or Other; p = 0.7859, Mixed Models Repeated Measures; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.72 to 0.55]
Statistical Analysis 2: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 1; Test type: Superiority or Other; p = 0.6429, Mixed Models Repeated Measures; Median Difference (Final Values) = -0.15, 95% CI 2-sided [-0.79 to 0.49]
Statistical Analysis 3: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 2; Test type: Superiority or Other; p = 0.0092, Mixed Models Repeated Measures; Mean Difference (Net) = -1.04, 95% CI 2-sided [-1.82 to -0.26]
Statistical Analysis 4: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 2; Test type: Superiority or Other; p = 0.0230, Mixed Models Repeated Measures; Mean Difference (Net) = -0.91, 95% CI 2-sided [-1.69 to -0.13]
Statistical Analysis 5: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 4; Test type: Superiority or Other; p = 0.0104, Mixed Models Repeated Measures; Mean Difference (Net) = -1.29, 95% CI 2-sided [-2.27 to -0.31]
Statistical Analysis 6: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 4; Test type: Superiority or Other; p = 0.0010, Mixed Models Repeated Measures; Mean Difference (Net) = -1.68, 95% CI 2-sided [-2.67 to -0.69]
Statistical Analysis 7: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 6; Test type: Superiority or Other; p = 0.0361, Mixed Models Repeated Measures; Mean Difference (Net) = -1.22, 95% CI 2-sided [-2.37 to -0.08]
Statistical Analysis 8: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 6; Test type: Superiority or Other; p = 0.0092, Mixed Models Repeated Measures; Mean Difference (Net) = -1.54, 95% CI [-2.69 to -0.38]

5. Secondary Outcome: Change From Baseline in the 16-item Quick Inventory of Depressive Symptomatology (QIDS-SR 16) Total Score
Description: The QIDS-SR is a self-report rating scale that assesses symptom severity of major depressive disorders. The QIDS-SR utilized during this study contained 16 separate items which correspond to 9 symptom criterion domains: (1) sad mood, (2) concentration, (3) self-criticism, (4) suicidal ideation,(5) interest, (6) energy/fatigue, (7) sleep disturbance (initial, middle, and late insomnia or hypersomnia), (8) decrease/increase in appetite/weight, and (9) psychomotor agitation/retardation. The QIDS-SR total score was calculated using the sum of the domain scores. The highest possible total QIDS-SR score is 27, which represents the most severe measure of depression. The lowest possible score is 0, which represents an absence of depression. Baseline was Day 1. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Day 1) to Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | Orvepitant 30 mg | Orvepitant 60 mg
Number analyzed (Participants) | 103 | 110 | 107
Scores on a Scale
  Week 1: number analyzed (Participants) | 102 | 109 | 103
  Week 1 | -2.47 (0.381) | -3.19 (0.364) | -3.13 (0.375)
  Week 2: number analyzed (Participants) | 94 | 102 | 100
  Week 2 | -3.48 (0.428) | -4.50 (0.408) | -4.03 (0.415)
  Week 4: number analyzed (Participants) | 85 | 95 | 93
  Week 4 | -4.16 (0.483) | -5.85 (0.457) | -6.26 (0.466)
  Week 6: number analyzed (Participants) | 77 | 85 | 83
  Week 6 | -5.05 (0.551) | -6.34 (0.523) | -6.73 (0.532)
Statistical Analysis 1: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 1; Test type: Superiority or Other; p = 0.1662, Mixed Models Repeated Measures; Mean Difference (Net) = -0.72, 95% CI 2-sided [-1.74 to 0.30]
Statistical Analysis 2: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 1; Test type: Superiority or Other; p = 0.2116, Mixed Models Repeated Measures; Mean Difference (Net) = -0.66, 95% CI 2-sided [-1.69 to 0.38]
Statistical Analysis 3: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 2; Test type: Superiority or Other; p = 0.0820, Mixed Models Repeated Measures; Mean Difference (Net) = -1.02, 95% CI 2-sided [-2.17 to 0.13]
Statistical Analysis 4: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 2; Test type: Superiority or Other; p = 0.3498, Mixed Models Repeated Measures; Mean Difference (Net) = -0.55, 95% CI 2-sided [-1.71 to 0.61]
Statistical Analysis 5: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 4; Test type: Superiority or Other; p = 0.0107, Mixed Models Repeated Measures; Mean Difference (Net) = -1.69, 95% CI 2-sided [-2.99 to -0.40]
Statistical Analysis 6: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 4; Test type: Superiority or Other; p = 0.0017, Mixed Models Repeated Measures; Mean Difference (Net) = -2.10, 95% CI 2-sided [-3.40 to -0.79]
Statistical Analysis 7: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 6; Test type: Superiority or Other; p = 0.0880, Mixed Models Repeated Measures; Mean Difference (Net) = -1.29, 95% CI 2-sided [-2.78 to 0.19]
Statistical Analysis 8: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 6; Test type: Superiority or Other; p = 0.0282, Mixed Models Repeated Measures; Mean Difference (Net) = -1.68, 95% CI 2-sided [-3.17 to -0.18]

6. Secondary Outcome: Change From Baseline in the HAM-D Anxiety Factor Score (Sum of Items 10, 11, 12, 13, 15 and 17)
Description: The HAMD anxiety factor score includes 6 items/questions (item 10: anxiety psychic, item 11: anxiety somatic, item 12: somatic symptoms gastrointestinal, item 13: somatic symptoms general, item 15: hypochondriasis and item 17: insight). The items are rated on a scale of 0 to 4 (items 10, 11 and 15) or 0 to 2 (items 12, 13 and 17), higher scores reflecting greater severity. The highest possible score is 18, which represents the most severe measure of anxiety; the lowest possible score is 0, which represents an absence of anxiety. Baseline was Day 1. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Day 1) to Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | Orvepitant 30 mg | Orvepitant 60 mg
Number analyzed (Participants) | 103 | 110 | 107
Scores on a Scale
  Week 1: number analyzed (Participants) | 102 | 110 | 103
  Week 1 | -1.06 (0.165) | -1.07 (0.157) | -1.28 (0.163)
  Week 2: number analyzed (Participants) | 94 | 102 | 100
  Week 2 | -1.47 (0.188) | -1.90 (0.179) | -1.91 (0.183)
  Week 4: number analyzed (Participants) | 85 | 97 | 93
  Week 4 | -2.19 (0.226) | -2.51 (0.212) | -2.78 (0.218)
  Week 6: number analyzed (Participants) | 78 | 86 | 84
  Week 6 | -2.60 (0.256) | -3.06 (0.242) | -3.30 (0.248)
Statistical Analysis 1: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 1; Test type: Superiority or Other; p = 0.9854, Mixed Models Repeated Measures; Mean Difference (Net) = -0.00, 95% CI 2-sided [-0.45 to 0.44]
Statistical Analysis 2: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 1; Test type: Superiority or Other; p = 0.3476, Mixed Models Repeated Measures; Mean Difference (Net) = -0.21, 95% CI 2-sided [-0.66 to 0.23]
Statistical Analysis 3: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 2; Test type: Superiority or Other; p = 0.0898, Mixed Models Repeated Measures; Mean Difference (Net) = -0.44, 95% CI 2-sided [-0.94 to 0.07]
Statistical Analysis 4: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 2; Test type: Superiority or Other; p = 0.0928, Mixed Models Repeated Measures; Mean Difference (Net) = -0.44, 95% CI 2-sided [-0.95 to 0.07]
Statistical Analysis 5: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 4; Test type: Superiority or Other; p = 0.2937, Mixed Models Repeated Measures; Mean Difference (Net) = -0.32, 95% CI 2-sided [-0.93 to 0.28]
Statistical Analysis 6: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 4; Test type: Superiority or Other; p = 0.0587, Mixed Models Repeated Measures; Mean Difference (Net) = -0.59, 95% CI 2-sided [-1.20 to 0.02]
Statistical Analysis 7: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 6; Test type: Superiority or Other; p = 0.1950, Mixed Models Repeated Measures; Mean Difference (Net) = -0.45, 95% CI 2-sided [-1.14 to 0.23]
Statistical Analysis 8: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 6; Test type: Superiority or Other; p = 0.0498, Mixed Models Repeated Measures; Mean Difference (Net) = -0.70, 95% CI 2-sided [-1.40 to -0.00]

7. Secondary Outcome: Percentage of Participants With Clinical Global Impression- Global Improvement (CGI-I) Score of 1 (Very Much Improved) or 2 (Much Improved)
Description: The CGI is a widely accepted measure of illness severity and clinical improvement in a variety of psychiatric disorders. Global improvement (CGI-I) item is rated on a 1-7 scale. The CGI-I assessed scores range from 1 - very much improved to 7 - very much worse. For the CGI-I, the investigator or delegated qualified clinician indicated their assessment of the participant's total improvement or worsening compared with the individual's condition at the start of the study whether or not the change was judged to be due to drug treatment. A participant with a CGI-I score of 1 'very much improved' or 2 'much improved' was considered a responder. Percentage of responders are reported.
Time Frame: Up to Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Orvepitant 30 mg | Orvepitant 60 mg
Number analyzed (Participants) | 103 | 110 | 107
Percentage of participants
  Week 1: number analyzed (Participants) | 102 | 110 | 103
  Week 1 | 5 | 10 | 4
  Week 2: number analyzed (Participants) | 94 | 102 | 100
  Week 2 | 10 | 22 | 16
  Week 4: number analyzed (Participants) | 85 | 97 | 93
  Week 4 | 22 | 35 | 32
  Week 6: number analyzed (Participants) | 78 | 86 | 84
  Week 6 | 31 | 44 | 40
Statistical Analysis 1: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 1; Test type: Superiority or Other; p = 0.1731, Regression, Logistic; Adjusted Odds Ratio = 2.14, 95% CI 2-sided [0.72 to 6.40]
Statistical Analysis 2: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 1; Test type: Superiority or Other; p = 0.7084, Regression, Logistic; Adjusted Odds Ratio = 0.77, 95% CI 2-sided [0.20 to 2.97]
Statistical Analysis 3: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 2; Test type: Superiority or Other; p = 0.0247, Regression, Logistic; Adjusted Odds Ratio = 2.60, 95% CI 2-sided [1.13 to 5.98]
Statistical Analysis 4: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 2; Test type: Superiority or Other; p = 0.1862, Regression, Logistic; Adjusted Odds Ratio = 1.80, 95% CI 2-sided [0.75 to 4.30]
Statistical Analysis 5: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 4; Test type: Superiority or Other; p = 0.0630, Regression, Logistic; Adjusted Odds Ratio = 1.87, 95% CI 2-sided [0.97 to 3.61]
Statistical Analysis 6: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 4; Test type: Superiority or Other; p = 0.1413, Regression, Logistic; Adjusted Odds Ratio = 1.65, 95% CI 2-sided [0.85 to 3.23]
Statistical Analysis 7: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 6; Test type: Superiority or Other; p = 0.0806, Regression, Logistic; Adjusted Odds Ratio = 1.77, 95% CI 2-sided [0.93 to 3.37]
Statistical Analysis 8: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 6; Test type: Superiority or Other; p = 0.2007, Regression, Logistic; Adjusted Odds Ratio = 1.53, 95% CI 2-sided [0.80 to 2.92]

8. Secondary Outcome: Change From Baseline in the Clinical Global Impression-Severity of Illness (CGI-S) Score
Description: The CGI is a widely accepted measure of illness severity and clinical improvement in a variety of psychiatric disorders. For the CGI-S, an independent site rater assessed the participant's severity of illness considering (1) their total clinical experience with the particular population being studied and (2) information obtained during the Baseline HAM-D interview with the participant. The severity of illness (CGI-S) item is rated on a 1 to 7 scale such that 1 (normal, not at all ill) and 7 (among the most extremely ill). Higher scores indicate worsening. Baseline was Day 1. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Day 1) to Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | Orvepitant 30 mg | Orvepitant 60 mg
Number analyzed (Participants) | 103 | 110 | 107
Scores on a Scale
  Week 1: number analyzed (Participants) | 102 | 110 | 103
  Week 1 | -0.34 (0.060) | -0.43 (0.057) | -0.43 (0.059)
  Week 2: number analyzed (Participants) | 94 | 102 | 100
  Week 2 | -0.51 (0.077) | -0.88 (0.073) | -0.73 (0.074)
  Week 4: number analyzed (Participants) | 85 | 97 | 93
  Week 4 | -0.80 (0.104) | -1.14 (0.098) | -1.26 (0.100)
  Week 6: number analyzed (Participants) | 78 | 86 | 84
  Week 6 | -1.07 (0.127) | -1.52 (0.120) | -1.56 (0.122)
Statistical Analysis 1: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 1; Test type: Superiority or Other; p = 0.2523, Mixed Models Repeated Measures; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.25 to 0.07]
Statistical Analysis 2: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 1; Test type: Superiority or Other; p = 0.2639, Mixed Models Repeated Measures; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.25 to 0.07]
Statistical Analysis 3: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 2; Test type: Superiority or Other; p = 0.0004, Mixed Models Repeated Measures; Mean Difference (Net) = -0.37, 95% CI 2-sided [-0.58 to -0.17]
Statistical Analysis 4: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 2; Test type: Superiority or Other; p = 0.0348, Mixed Models Repeated Measures; Mean Difference (Net) = -0.22, 95% CI 2-sided [-0.43 to -0.02]
Statistical Analysis 5: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 4; Test type: Superiority or Other; p = 0.0166, Mixed Models Repeated Measures; Mean Difference (Net) = -0.34, 95% CI 2-sided [-0.62 to -0.06]
Statistical Analysis 6: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 4; Test type: Superiority or Other; p = 0.0014, Mixed Models Repeated Measures; Mean Difference (Net) = -0.46, 95% CI 2-sided [-0.75 to -0.18]
Statistical Analysis 7: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 6; Test type: Superiority or Other; p = 0.0099, Mixed Models Repeated Measures; Mean Difference (Net) = -0.45, 95% CI 2-sided [-0.79 to -0.11]
Statistical Analysis 8: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 6; Test type: Superiority or Other; p = 0.0059, Mixed Models Repeated Measures; Mean Difference (Net) = -0.49, 95% CI 2-sided [-0.83 to -0.14]

9. Secondary Outcome: Change From Baseline in the Cognitive and Physical Function Questionnaire (CPFQ) Total Score
Description: The CPFQ is a brief self-report scale which is designed to measure cognitive and executive dysfunction in mood and anxiety disorders. The scale comprises 7 questions assessing each of the most common complaints of depressed participants reporting fatigue or cognitive/executive problems. Each question is rated on a scale of 1 to 6, (1 = greater than normal; 2 = normal; 3 = minimally diminished; 4=moderately diminished; 5 = markedly diminished; and 6 = totally absent). The following five areas were included: motivation/interest/enthusiasm; wakefulness/alertness; energy; focus/sustain attention; remember/recall information; find words and sharpness/mental acuity. The total score (sum of individual question scores) ranged from 7 to 42. Lower score 7 represents greater than normal functioning and higher score 42 indicate poorer functioning (worst outcome). Baseline was Day 1. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Day 1) and Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | Orvepitant 30 mg | Orvepitant 60 mg
Number analyzed (Participants) | 103 | 110 | 107
Scores on a Scale
  Week 1: number analyzed (Participants) | 101 | 109 | 103
  Week 1 | -3.24 (0.582) | -3.72 (0.553) | -3.22 (0.572)
  Week 2: number analyzed (Participants) | 94 | 100 | 100
  Week 2 | -3.80 (0.567) | -5.31 (0.541) | -4.37 (0.550)
  Week 4: number analyzed (Participants) | 85 | 94 | 92
  Week 4 | -5.12 (0.659) | -6.34 (0.623) | -6.27 (0.637)
  Week 6: number analyzed (Participants) | 78 | 84 | 84
  Week 6 | -5.51 (0.729) | -7.67 (0.693) | -7.85 (0.704)
Statistical Analysis 1: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 1; Test type: Superiority or Other; p = 0.5473, Mixed Models Repeated Measures; Mean Difference (Net) = -0.48, 95% CI 2-sided [-2.04 to 1.08]
Statistical Analysis 2: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 1; Test type: Superiority or Other; p = 0.9814, Mixed Models Repeated Measures; Mean Difference (Net) = 0.02, 95% CI 2-sided [-1.56 to 1.60]
Statistical Analysis 3: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 2; Test type: Superiority or Other; p = 0.0515, Mixed Models Repeated Measures; Mean Difference (Net) = -1.51, 95% CI 2-sided [-3.03 to 0.01]
Statistical Analysis 4: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 2; Test type: Superiority or Other; p = 0.4680, Mixed Models Repeated Measures; Mean Difference (Net) = -0.56, 95% CI 2-sided [-2.09 to 0.96]
Statistical Analysis 5: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 4; Test type: Superiority or Other; p = 0.1757, Mixed Models Repeated Measures; Mean Difference (Net) = -1.22, 95% CI 2-sided [-2.98 to 0.55]
Statistical Analysis 6: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 4; Test type: Superiority or Other; p = 0.2048, Mixed Models Repeated Measures; Mean Difference (Net) = -1.15, 95% CI 2-sided [-2.93 to 0.63]
Statistical Analysis 7: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 6; Test type: Superiority or Other; p = 0.0312, Mixed Models Repeated Measures; Mean Difference (Net) = -2.16, 95% CI 2-sided [-4.12 to -0.20]
Statistical Analysis 8: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 6; Test type: Superiority or Other; p = 0.0202, Mixed Models Repeated Measures; Mean Difference (Net) = -2.34, 95% CI 2-sided [-4.31 to -0.37]

10. Secondary Outcome: Change From Baseline in Morning Sleep Questionnaire (MSQ) Values for Total Sleep Time (TST), Sleep Onset Latency (SOL) and Wake Time After Sleep Onset (WTSO)
Description: The MSQ is a self-rated scale designed to assess effects on sleep and effects on next day functioning. The following six variables were assessed in order to determine effects on sleep: (1) total sleep time, (2) sleep onset latency, (3) number of nocturnal awakenings, (4) wake time after sleep onset, (5) sleep quality (where poor=1 and excellent= 10) and (6) the refreshing value of the sleep (where poor=1 and excellent= 10). During the conduct of the study, participants self-administered the MSQ via an Interactive Voice Response System (IVRS) from their home the morning of each clinic visit. Participants were provided paper MSQ diary cards for note taking prior to completing the IVRS call. If a participant did not remember to place the IVRS MSQ call the morning of the clinic visit from home, they were allowed to place the call during in the clinic during their visit. Baseline was Day 1. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Day 1) to Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Minutes (mins)
Arm/Group | Placebo | Orvepitant 30 mg | Orvepitant 60 mg
Number analyzed (Participants) | 103 | 110 | 107
Minutes (mins)
  TST; Week 1 | 36.09 (9.204) | 40.54 (8.834) | 63.46 (9.148)
  TST; Week 2 | 34.62 (9.728) | 42.74 (9.371) | 48.14 (9.440)
  TST; Week 4 | 49.57 (10.991) | 32.07 (10.309) | 70.68 (10.472)
  TST; Week 6 | 39.79 (9.930) | 44.26 (9.443) | 51.26 (9.523)
  SOL; Week 1 | -7.16 (5.658) | -18.68 (5.440) | -31.06 (5.620)
  SOL; Week 2 | -14.60 (5.609) | -22.27 (5.405) | -39.28 (5.444)
  SOL; Week 4 | -21.75 (6.354) | -32.46 (5.949) | -37.06 (6.041)
  SOL; Week 6 | -34.50 (5.212) | -27.66 (4.940) | -37.75 (4.998)
  WTSO; Week 1 | -12.09 (7.248) | -9.69 (6.799) | -21.38 (7.252)
  WTSO; Week 2 | -2.12 (7.397) | -17.99 (7.196) | -24.38 (7.343)
  WTSO; Week 4 | -15.76 (11.019) | -13.60 (10.306) | -17.43 (10.819)
  WTSO; Week 6 | -16.99 (10.713) | -21.08 (10.428) | -14.08 (11.198)
Statistical Analysis 1: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg, TST at Week 1; Test type: Superiority or Other; p = 0.7246, Mixed Models Repeated Measures; Mean Difference (Net) = 4.45, 95% CI 2-sided [-20.38 to 29.28]
Statistical Analysis 2: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg, TST at Week 1; Test type: Superiority or Other; p = 0.0332, Mixed Models Repeated Measures; Mean Difference (Net) = 27.36, 95% CI 2-sided [2.20 to 52.52]
Statistical Analysis 3: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg, TST at Week 2; Test type: Superiority or Other; p = 0.5439, Mixed Models Repeated Measures; Mean Difference (Net) = 8.12, 95% CI 2-sided [-18.18 to 34.41]
Statistical Analysis 4: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg, TST at Week 2; Test type: Superiority or Other; p = 0.3127, Mixed Models Repeated Measures; Mean Difference (Net) = 13.52, 95% CI 2-sided [-12.80 to 39.85]
Statistical Analysis 5: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg, TST at Week 4; Test type: Superiority or Other; p = 0.2419, Mixed Models Repeated Measures; Mean Difference (Net) = -17.51, 95% CI 2-sided [-46.90 to 11.89]
Statistical Analysis 6: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg, TST at Week 4; Test type: Superiority or Other; p = 0.1606, Mixed Models Repeated Measures; Median Difference (Net) = 21.11, 95% CI 2-sided [-8.43 to 50.64]
Statistical Analysis 7: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg, TST at Week 6; Test type: Superiority or Other; p = 0.7412, Mixed Models Repeated Measures; Mean Difference (Net) = 4.48, 95% CI [-22.21 to 31.16]
Statistical Analysis 8: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg, TST at Week 6; Test type: Superiority or Other; p = 0.3974, Mixed Models Repeated Measures; Mean Difference (Final Values) = 11.47, 95% CI 2-sided [-15.19 to 38.14]
Statistical Analysis 9: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg, SOL at Week 1; Test type: Superiority or Other; p = 0.1397, Mixed Models Repeated Measures; Mean Difference (Net) = -11.52, 95% CI 2-sided [-26.83 to 3.79]
Statistical Analysis 10: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg, SOL at Week 1; Test type: Superiority or Other; p = 0.0026, Mixed Models Repeated Measures; Mean Difference (Net) = -23.90, 95% CI 2-sided [-39.40 to -8.41]
Statistical Analysis 11: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg, SOL at Week 2; Test type: Superiority or Other; p = 0.3206, Mixed Models Repeated Measures; Mean Difference (Net) = -7.67, 95% CI 2-sided [-22.85 to 7.50]
Statistical Analysis 12: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg, SOL at Week 2; Test type: Superiority or Other; p = 0.0015, Mixed Models Repeated Measures; Mean Difference (Net) = -24.67, 95% CI 2-sided [-39.86 to -9.49]
Statistical Analysis 13: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg, SOL at Week 4; Test type: Superiority or Other; p = 0.2157, Mixed Models Repeated Measures; Mean Difference (Net) = -10.71, 95% CI 2-sided [-27.70 to 6.28]
Statistical Analysis 14: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg, SOL at Week 4; Test type: Superiority or Other; p = 0.0784, Mixed Models Repeated Measures; Mean Difference (Net) = -15.31, 95% CI 2-sided [-32.37 to 1.75]
Statistical Analysis 15: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg, SOL at Week 6; Test type: Superiority or Other; p = 0.3345, Mixed Models Repeated Measures; Mean Difference (Net) = 6.84, 95% CI 2-sided [-7.09 to 20.78]
Statistical Analysis 16: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg, SOL at Week 6; Test type: Superiority or Other; p = 0.6471, Mixed Models Repeated Measures; Mean Difference (Net) = -3.25, 95% CI 2-sided [-17.19 to 10.70]
Statistical Analysis 17: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg, WTSO at Week 1; Test type: Superiority or Other; p = 0.8071, Mixed Models Repeated Measures; Mean Difference (Net) = 2.40, 95% CI 2-sided [-16.95 to 21.75]
Statistical Analysis 18: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg, WTSO at Week 1; Test type: Superiority or Other; p = 0.3564, Mixed Models Repeated Measures; Mean Difference (Net) = -9.30, 95% CI 2-sided [-29.11 to 10.52]
Statistical Analysis 19: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg, WTSO at Week 2; Test type: Superiority or Other; p = 0.1220, Mixed Models Repeated Measures; Mean Difference (Net) = -15.86, 95% CI 2-sided [-36.00 to 4.28]
Statistical Analysis 20: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg, WTSO at Week 2; Test type: Superiority or Other; p = 0.0313, Mixed Models Repeated Measures; Mean Difference (Net) = -22.25, 95% CI 2-sided [-42.49 to -2.01]
Statistical Analysis 21: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg, WTSO at Week 4; Test type: Superiority or Other; p = 0.8861, Mixed Models Repeated Measures; Mean Difference (Net) = 2.15, 95% CI 2-sided [-27.45 to 31.76]
Statistical Analysis 22: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg, WTSO at Week 4; Test type: Superiority or Other; p = 0.9132, Mixed Models Repeated Measures; Mean Difference (Net) = -1.67, 95% CI 2-sided [-31.87 to 28.53]
Statistical Analysis 23: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg, WTSO at Week 6; Test type: Superiority or Other; p = 0.7844, Mixed Models Repeated Measures; Mean Difference (Net) = -4.09, 95% CI 2-sided [-33.55 to 25.37]
Statistical Analysis 24: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 30 mg, WTSO at Week 6; Test type: Superiority or Other; p = 0.8497, Mixed Models Repeated Measures; Mean Difference (Net) = 2.90, 95% CI 2-sided [-27.33 to 33.14]

11. Secondary Outcome: Change From Baseline in MSQ Values for Number of Nocturnal Awakenings
Description: as for outcome 10
Time Frame: Baseline (Day 1) to Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Awakenings
Arm/Group | Placebo | Orvepitant 30 mg | Orvepitant 60 mg
Number analyzed (Participants) | 103 | 110 | 107
Awakenings
  Week 1: number analyzed (Participants) | 73 | 80 | 72
  Week 1 | -0.07 (0.225) | -0.29 (0.214) | 0.09 (0.227)
  Week 2: number analyzed (Participants) | 68 | 69 | 68
  Week 2 | -0.42 (0.120) | -0.53 (0.116) | -0.66 (0.119)
  Week 4: number analyzed (Participants) | 55 | 61 | 58
  Week 4 | -0.42 (0.140) | -0.41 (0.130) | -0.71 (0.137)
  Week 6: number analyzed (Participants) | 50 | 51 | 46
  Week 6 | -0.36 (0.152) | -0.67 (0.147) | -0.84 (0.157)
Statistical Analysis 1: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 1; Test type: Superiority or Other; p = 0.4814, Mixed Models Repeated Measures; Mean Difference (Net) = -0.22, 95% CI 2-sided [-0.83 to 0.39]
Statistical Analysis 2: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 1; Test type: Superiority or Other; p = 0.6179, Mixed Models Repeated Measures; Mean Difference (Net) = 0.16, 95% CI 2-sided [-0.47 to 0.79]
Statistical Analysis 3: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 2; Test type: Superiority or Other; p = 0.5022, Mixed Models Repeated Measures; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.44 to 0.21]
Statistical Analysis 4: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 2; Test type: Superiority or Other; p = 0.1389, Mixed Models Repeated Measures; Mean Difference (Net) = -0.25, 95% CI 2-sided [-0.57 to 0.08]
Statistical Analysis 5: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 4; Test type: Superiority or Other; p = 0.9663, Mixed Models Repeated Measures; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.36 to 0.38]
Statistical Analysis 6: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 4; Test type: Superiority or Other; p = 0.1311, Mixed Models Repeated Measures; Mean Difference (Net) = -0.29, 95% CI 2-sided [-0.67 to 0.09]
Statistical Analysis 7: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 6; Test type: Superiority or Other; p = 0.1362, Mixed Models Repeated Measures; Mean Difference (Net) = -0.31, 95% CI 2-sided [-0.73 to 0.10]
Statistical Analysis 8: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 6; Test type: Superiority or Other; p = 0.0275, Mixed Models Repeated Measures; Mean Difference (Net) = -0.48, 95% CI 2-sided [-0.91 to -0.05]

12. Secondary Outcome: Change From Baseline in MSQ Values for Sleep Quality (SQ) and Refreshing Value of Sleep (RVS)
Description: The MSQ is a self-rated scale designed to assess effects on sleep and effects on next day functioning. The score relating to SQ and RVS was measured by items/questions 4 and 5 respectively of the MSQ. The following two variables SQ and RVS were assessed in order to determine effects on sleep. Participants were asked to rate their SQ and RVS on a scale of 1 to 10. This scale has no subscales. The total score for SQ and RVS, both, ranged from 1 to 10 where 1=poor and 10=excellent. Lower scores indicated poor SQ and RVS and higher scores indicated excellent SQ and excellent RVS. During the conduct of study, participants self-administered MSQ via an IVRS from their home the morning of each clinic visit. If a participant did not remember to place IVRS MSQ call the morning of the clinic visit from home, they were allowed to place call during in the clinic during their visit. Baseline was Day 1. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Day 1) to Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | Orvepitant 30 mg | Orvepitant 60 mg
Number analyzed (Participants) | 103 | 110 | 107
Scores on a Scale
  SQ; Week 1: number analyzed (Participants) | 99 | 105 | 99
  SQ; Week 1 | 0.79 (0.201) | 1.30 (0.192) | 1.48 (0.199)
  SQ; Week 2: number analyzed (Participants) | 92 | 97 | 97
  SQ; Week 2 | 0.81 (0.207) | 1.75 (0.199) | 1.65 (0.201)
  SQ; Week 4: number analyzed (Participants) | 83 | 94 | 92
  SQ; Week 4 | 1.45 (0.224) | 1.58 (0.209) | 2.27 (0.214)
  SQ; Week 6: number analyzed (Participants) | 76 | 83 | 83
  SQ; Week 6 | 1.53 (0.238) | 2.19 (0.226) | 2.30 (0.228)
  RVS; Week 1: number analyzed (Participants) | 99 | 105 | 99
  RVS; Week 1 | 0.75 (0.198) | 1.14 (0.190) | 1.45 (0.196)
  RVS; Week 2: number analyzed (Participants) | 92 | 97 | 97
  RVS; Week 2 | 1.10 (0.208) | 1.70 (0.200) | 1.69 (0.202)
  RVS; Week 4: number analyzed (Participants) | 83 | 94 | 92
  RVS; Week 4 | 1.55 (0.230) | 1.52 (0.215) | 2.32 (0.219)
  RVS; Week 6: number analyzed (Participants) | 76 | 83 | 83
  RVS; Week 6 | 1.67 (0.246) | 2.31 (0.234) | 2.41 (0.236)
Statistical Analysis 1: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg, SQ at Week 1; Test type: Superiority or Other; p = 0.0606, Mixed Models Repeated Measures; Mean Difference (Net) = 0.52, 95% CI 2-sided [-0.02 to 1.06]
Statistical Analysis 2: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg, SQ at Week 1; Test type: Superiority or Other; p = 0.0132, Mixed Models Repeated Measures; Mean Difference (Net) = 0.69, 95% CI 2-sided [0.15 to 1.24]
Statistical Analysis 3: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg, SQ at Week 2; Test type: Superiority or Other; p = 0.0010, Mixed Models Repeated Measures; Mean Difference (Net) = 0.94, 95% CI 2-sided [0.38 to 1.50]
Statistical Analysis 4: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg, SQ at Week 2; Test type: Superiority or Other; p = 0.0034, Mixed Models Repeated Measures; Mean Difference (Net) = 0.84, 95% CI 2-sided [0.28 to 1.40]
Statistical Analysis 5: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg, SQ at Week 4; Test type: Superiority or Other; p = 0.6692, Mixed Models Repeated Measures; Mean Difference (Net) = 0.13, 95% CI 2-sided [-0.47 to 0.72]
Statistical Analysis 6: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg, SQ at Week 4; Test type: Superiority or Other; p = 0.0078, Mixed Models Repeated Measures; Mean Difference (Net) = 0.82, 95% CI 2-sided [0.22 to 1.42]
Statistical Analysis 7: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg, SQ at Week 6; Test type: Superiority or Other; p = 0.0440, Mixed Models Repeated Measures; Mean Difference (Net) = 0.66, 95% CI 2-sided [0.02 to 1.30]
Statistical Analysis 8: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg, SQ at Week 6; Test type: Superiority or Other; p = 0.0181, Mixed Models Repeated Measures; Mean Difference (Net) = 0.77, 95% CI 2-sided [0.13 to 1.41]
Statistical Analysis 9: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg, RVS at Week 1; Test type: Superiority or Other; p = 0.1484, Mixed Models Repeated Measures; Mean Difference (Net) = 0.39, 95% CI 2-sided [-0.14 to 0.92]
Statistical Analysis 10: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg, RVS at Week 1; Test type: Superiority or Other; p = 0.0108, Mixed Models Repeated Measures; Mean Difference (Net) = 0.70, 95% CI 2-sided [0.16 to 1.24]
Statistical Analysis 11: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg, RVS at Week 2; Test type: Superiority or Other; p = 0.0361, Mixed Models Repeated Measures; Mean Difference (Net) = 0.60, 95% CI [0.04 to 1.16]
Statistical Analysis 12: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg, RVS at Week 2; Test type: Superiority or Other; p = 0.0418, Mixed Models Repeated Measures; Mean Difference (Net) = 0.58, 95% CI 2-sided [0.02 to 1.15]
Statistical Analysis 13: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg, RVS at Week 4; Test type: Superiority or Other; p = 0.9305, Mixed Models Repeated Measures; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.64 to 0.58]
Statistical Analysis 14: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg, RVS at Week 4; Test type: Superiority or Other; p = 0.0141, Mixed Models Repeated Measures; Mean Difference (Net) = 0.77, 95% CI 2-sided [0.16 to 1.39]
Statistical Analysis 15: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg, RVS at Week 6; Test type: Superiority or Other; p = 0.0562, Mixed Models Repeated Measures; Mean Difference (Net) = 0.65, 95% CI 2-sided [-0.02 to 1.31]
Statistical Analysis 16: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 30 mg, RVS at Week 6; Test type: Superiority or Other; p = 0.0296, Mixed Models Repeated Measures; Mean Difference (Net) = 0.74, 95% CI 2-sided [0.07 to 1.40]

13. Secondary Outcome: Number of Participants Who Remit (Have an Endpoint HAM-D Total Score <= 7) Who Continue to Show Symptoms on the HAM-D Sleep Items
Description: A HAM-D remitter was defined as a participant with a HAM-D total score less than or equal to 7. The HAM-D was designed to measure the severity of depressive symptoms in participants with primary depressive illness. The scale is a checklist of items that are ranked on a scale of 0 to 4 or 0 to 2. Items with quantifiable severity are scored 0 to 4 (4 indicating the greatest severity) or 0 to 2 (2 indicating the greatest severity) with 0 indicating not present. The HAM-D Total Score is calculated by summing the individual response scores on the HAM-D questionnaire. The highest possible score is 52, which represents the most severe measure of depression; the lowest possible score is 0, which represents an absence of depression. The HAM-D is also useful for monitoring changes in depressive symptoms with treatment and in comparing the efficacy of various interventions if the participant requires more than one type of treatment.
Time Frame: Up to Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Orvepitant 30 mg | Orvepitant 60 mg
Number analyzed (Participants) | 103 | 110 | 107
Participants
  Week 1: number analyzed (Participants) | 102 | 110 | 103
  Week 1 | 1 | 2 | 0
  Week 2: number analyzed (Participants) | 94 | 102 | 100
  Week 2 | 2 | 2 | 4
  Week 4: number analyzed (Participants) | 85 | 97 | 93
  Week 4 | 5 | 10 | 10
  Week 6: number analyzed (Participants) | 78 | 86 | 84
  Week 6 | 8 | 16 | 15

14. Secondary Outcome: Number of Participants With Suicidal Behavior, Ideation, and Most Common Ideation Using the Columbia Suicidality Severity Rating Scale (C-SSRS)
Description: The C-SSRS is a clinician-rated scale that evaluates severity and change of suicidality by integrating both behavior and ideation. It has 3 sections, Suicidal Behavior (SB), Suicidal Ideation (SI) and Intensity of Ideation (II). For SB, participants (par) were scored non-suicidal:0, preparatory acts or behavior communicating ideation:1, aborted attempt:2, interrupted attempt:3 or actual attempt:4 (most severe). For SI, par were scored non-suicidal:0, wish to be dead:1, non-specific active suicidal thoughts:2, active suicidal ideation with associated thoughts of methods without intent:3, active suicidal ideation with some intent to act on suicidal thoughts without clear plan:4, active suicidal ideation with plan and intent:5 (most severe). II scale made of 5 questions measuring frequency, duration, controllability, deterrent and reasons; par received a separate score on most common ideation and on most severe. Total II score is obtained by adding scores from all 5 questions.
Time Frame: Week 8
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Orvepitant 30 mg | Orvepitant 60 mg
Number analyzed (Participants) | 103 | 110 | 107
Participants
  Suicidal Ideation score 1 | 27 | 26 | 27
  Suicidal Ideation score 2 | 5 | 7 | 6
  Suicidal Ideation score 3 | 1 | 3 | 4
  Suicidal Ideation score 4 | 0 | 1 | 0
  Suicidal Ideation score 5 | 1 | 1 | 0

15. Secondary Outcome: Number of Discontinuation-emergent Signs and Symptoms Using the Discontinuation-Emergent Signs and Symptoms (DESS)
Description: The discontinuation signs and symptoms scale consists of 43 signs and symptoms, scored as 'new symptom', 'old symptom but worse', 'old symptom but improved' or ' symptom not present/old symptom but unchanged'. A frequency table for each symptom is reported by treatment and visit. The total number of new signs and symptoms, old symptoms but worse, old symptoms but improved and the total number of new or old-but-worse signs and symptoms are calculated for treatment and visit and reported.
Time Frame: Week 1 to Week 8/Follow up 1
Population: All subjects population comprised of all participants who received at least one dose of study medication. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Signs and symptoms
Arm/Group | Placebo | Orvepitant 30 mg | Orvepitant 60 mg
Number analyzed (Participants) | 108 | 113 | 107
Signs and symptoms
  New symptom; Week 1: number analyzed (Participants) | 2 | 1 | 1
  New symptom; Week 1 | 1.5 (0.71) | 2.0 (NA) — Single participant analyzed | 2.0 (NA) — Single participant analyzed
  Old Symptom But Improved; Week 1: number analyzed (Participants) | 1 | 0 | 1
  Old Symptom But Improved; Week 1 | 1.0 (NA) — Single participant |  | 3.0 (NA) — Single participant
  Old Symptom But Worsened; Week 1: number analyzed (Participants) | 3 | 0 | 3
  Old Symptom But Worsened; Week 1 | 5.7 (4.04) |  | 1.0 (0.00)
  Unchanged/ Not present; Week 1: number analyzed (Participants) | 6 | 5 | 4
  Unchanged/ Not present; Week 1 | 39.5 (5.09) | 42.6 (0.89) | 41.0 (2.71)
  New or Old but Worsened; Week 1: number analyzed (Participants) | 3 | 1 | 3
  New or Old but Worsened; Week 1 | 6.7 (4.93) | 2.0 (NA) — Single participant analyzed | 1.7 (1.15)
  New symptom; Week 2: number analyzed (Participants) | 0 | 1 | 0
  New symptom; Week 2 |  | 1.0 (NA) — Single participant analyzed |
  Old Symptom But Improved; Week 2: number analyzed (Participants) | 0 | 3 | 0
  Old Symptom But Improved; Week 2 |  | 3.0 (3.46) |
  Old Symptom But Worsened; Week 2: number analyzed (Participants) | 0 | 0 | 2
  Old Symptom But Worsened; Week 2 |  |  | 6.0 (1.41)
  Unchanged/ Not present; Week 2: number analyzed (Participants) | 2 | 3 | 6
  Unchanged/ Not present; Week 2 | 43.0 (0.00) | 39.7 (3.21) | 41.0 (3.16)
  New or Old but Worsened; Week 2: number analyzed (Participants) | 0 | 1 | 2
  New or Old but Worsened; Week 2 |  | 1.0 (NA) — Single participant analyzed | 6.0 (1.41)
  New symptom; Week 4: number analyzed (Participants) | 1 | 2 | 2
  New symptom; Week 4 | 8.0 (NA) — Single participant analyzed | 1.5 (0.71) | 6.0 (5.66)
  Old Symptom But Improved; Week 4: number analyzed (Participants) | 2 | 3 | 2
  Old Symptom But Improved; Week 4 | 2.5 (0.71) | 4.7 (1.53) | 2.0 (1.41)
  Old Symptom But Worsened; Week 4: number analyzed (Participants) | 3 | 3 | 2
  Old Symptom But Worsened; Week 4 | 6.0 (4.36) | 11.7 (8.50) | 4.5 (0.71)
  Unchanged/ Not present; Week 4: number analyzed (Participants) | 9 | 10 | 6
  Unchanged/ Not present; Week 4 | 39.6 (4.98) | 37.8 (9.31) | 38.8 (6.82)
  New or Old but Worsened; Week 4: number analyzed (Participants) | 3 | 3 | 2
  New or Old but Worsened; Week 4 | 8.7 (4.93) | 12.7 (7.77) | 10.5 (6.36)
  New symptom; Week 6: number analyzed (Participants) | 8 | 21 | 15
  New symptom; Week 6 | 2.8 (3.45) | 2.1 (1.98) | 5.2 (7.74)
  Old Symptom But Improved; Week 6: number analyzed (Participants) | 24 | 39 | 40
  Old Symptom But Improved; Week 6 | 4.1 (2.98) | 4.0 (3.46) | 5.7 (7.41)
  Old Symptom But Worsened; Week 6: number analyzed (Participants) | 20 | 21 | 20
  Old Symptom But Worsened; Week 6 | 3.9 (3.75) | 2.7 (2.49) | 3.2 (3.15)
  Unchanged/ Not present; Week 6: number analyzed (Participants) | 78 | 85 | 83
  Unchanged/ Not present; Week 6 | 40.4 (3.82) | 40.0 (4.01) | 39.0 (6.48)
  New or Old but Worsened; Week 6: number analyzed (Participants) | 25 | 34 | 27
  New or Old but Worsened; Week 6 | 4.0 (3.82) | 3.0 (3.31) | 5.2 (7.01)
  New symptom; Follow-up 1: number analyzed (Participants) | 14 | 17 | 24
  New symptom; Follow-up 1 | 3.0 (3.37) | 1.8 (1.09) | 2.4 (1.86)
  Old Symptom But Improved; Follow-up 1: number analyzed (Participants) | 23 | 34 | 30
  Old Symptom But Improved; Follow-up 1 | 3.3 (2.43) | 2.6 (2.28) | 4.0 (2.58)
  Old Symptom But Worsened; Follow-up 1: number analyzed (Participants) | 18 | 29 | 25
  Old Symptom But Worsened; Follow-up 1 | 2.6 (1.82) | 3.9 (4.07) | 4.1 (3.72)
  Unchanged/ Not present; Follow-up 1: number analyzed (Participants) | 87 | 98 | 94
  Unchanged/ Not present; Follow-up 1 | 41.1 (3.65) | 40.6 (3.87) | 40.0 (4.25)
  New or Old but Worsened; Follow-up 1: number analyzed (Participants) | 20 | 36 | 33
  New or Old but Worsened; Follow-up 1 | 4.5 (4.22) | 4.0 (3.96) | 4.8 (4.01)

16. Secondary Outcome: Change From Baseline in the Massachusetts Sexual Function Questionnaire (MSFQ)-Males
Description: The MSFQ is a self report rating scale derived from the Guided Interview Questionnaire for females and males. The questionnaire includes five questions with a score for each question ranging from 1 to 6 (1 = greater than normal; 2 = normal; 3 = minimally diminished; 4=moderately diminished; 5 = markedly diminished; and 6 = totally absent). The following five areas of sexual functioning were included: (1) diminished/absent libido; (2) arousal difficulties; (3) orgasm difficulties/anorgasmia; (4) erectile dysfunction (males only) and (5) degree of sexual satisfaction. A total score (sum of individual question score) was used as a global measure of sexual dysfunction which ranged from 5 to 30, where 5 represents greater than normal functioning and 30 represents poorer function (worst outcome). Baseline was Day 1. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values. A negative change from Baseline was considered a positive outcome.
Time Frame: Baseline (Day 1) to Week 6
Population: Only males from all subjects population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | Orvepitant 30 mg | Orvepitant 60 mg
Number analyzed (Participants) | 32 | 45 | 37
Scores on a Scale
  Week 1: number analyzed (Participants) | 29 | 42 | 36
  Week 1 | -1.61 (0.961) | 0.58 (0.835) | -0.27 (0.894)
  Week 2: number analyzed (Participants) | 27 | 39 | 36
  Week 2 | -2.22 (1.050) | -1.16 (0.906) | -1.20 (0.952)
  Week 4: number analyzed (Participants) | 26 | 37 | 34
  Week 4 | -2.98 (1.080) | -1.49 (0.938) | -2.22 (0.983)
  Week 6: number analyzed (Participants) | 23 | 32 | 31
  Week 6 | -3.46 (1.168) | -2.25 (1.007) | -2.82 (1.046)
Statistical Analysis 1: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 1; Test type: Superiority or Other; p = 0.0735, Mixed Models Repeated Measures; Mean Difference (Net) = 2.20, 95% CI 2-sided [-0.21 to 4.61]
Statistical Analysis 2: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 1; Test type: Superiority or Other; p = 0.2905, Mixed Models Repeated Measures; Mean Difference (Net) = 1.35, 95% CI 2-sided [-1.17 to 3.86]
Statistical Analysis 3: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 2; Test type: Superiority or Other; p = 0.4327, Mixed Models Repeated Measures; Mean Difference (Net) = 1.05, 95% CI 2-sided [-1.60 to 3.70]
Statistical Analysis 4: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 2; Test type: Superiority or Other; p = 0.4642, Mixed Models Repeated Measures; Mean Difference (Net) = 1.01, 95% CI 2-sided [-1.73 to 3.75]
Statistical Analysis 5: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 4; Test type: Superiority or Other; p = 0.2850, Mixed Models Repeated Measures; Mean Difference (Net) = 1.48, 95% CI 2-sided [-1.26 to 4.23]
Statistical Analysis 6: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 4; Test type: Superiority or Other; p = 0.5984, Mixed Models Repeated Measures; Mean Difference (Net) = 0.75, 95% CI 2-sided [-2.08 to 3.59]
Statistical Analysis 7: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 6; Test type: Superiority or Other; p = 0.4192, Mixed Models Repeated Measures; Mean Difference (Net) = 1.21, 95% CI 2-sided [-1.76 to 4.19]
Statistical Analysis 8: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 6; Test type: Superiority or Other; p = 0.6766, Mixed Models Repeated Measures; Mean Difference (Net) = 0.64, 95% CI 2-sided [-2.42 to 3.71]

17. Secondary Outcome: Change From Baseline in the MSFQ Total Score-Females
Description: The MSFQ is a self report rating scale derived from the Guided Interview Questionnaire for females and males. The questionnaire includes five questions with a score for each question ranging from 1 to 6 (1 = greater than normal; 2 = normal; 3 = minimally diminished; 4=moderately diminished; 5 = markedly diminished; and 6 = totally absent). The following four areas of sexual functioning were included: (1) diminished/absent libido; (2) arousal difficulties; (3) orgasm difficulties/anorgasmia; and (4) degree of sexual satisfaction. A total score (sum of individual question score) was used as a global measure of sexual dysfunction which ranged from 4 to 24, where 5 represents greater than normal functioning and 24 represents poorer function (worst outcome). Baseline was Day 1. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values. A negative change from Baseline was considered a positive outcome.
Time Frame: Baseline (Day 1) to Week 6
Population: Only females from all subjects population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | Orvepitant 30 mg | Orvepitant 60 mg
Number analyzed (Participants) | 76 | 68 | 70
Scores on a Scale
  Week 1: number analyzed (Participants) | 71 | 68 | 67
  Week 1 | -0.76 (0.451) | -0.76 (0.455) | -0.67 (0.467)
  Week 2: number analyzed (Participants) | 66 | 63 | 64
  Week 2 | -1.30 (0.520) | -1.47 (0.526) | -0.70 (0.533)
  Week 4: number analyzed (Participants) | 59 | 58 | 59
  Week 4 | -2.31 (0.643) | -2.24 (0.641) | -2.89 (0.648)
  Week 6: number analyzed (Participants) | 54 | 53 | 52
  Week 6 | -2.13 (0.702) | -2.49 (0.697) | -4.40 (0.711)
Statistical Analysis 1: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 1; Test type: Superiority or Other; p = 0.9951, Mixed Models Repeated Measures; Mean Difference (Net) = -0.00, 95% CI 2-sided [-1.26 to 1.25]
Statistical Analysis 2: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 1; Test type: Superiority or Other; p = 0.8940, Mixed Models Repeated Measures; Mean Difference (Net) = 0.08, 95% CI 2-sided [-1.17 to 1.34]
Statistical Analysis 3: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 2; Test type: Superiority or Other; p = 0.8195, Mixed Models Repeated Measures; Mean Difference (Net) = -0.17, 95% CI 2-sided [-1.61 to 1.28]
Statistical Analysis 4: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 2; Test type: Superiority or Other; p = 0.4106, Mixed Models Repeated Measures; Mean Difference (Net) = 0.60, 95% CI 2-sided [-0.84 to 2.05]
Statistical Analysis 5: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 4; Test type: Superiority or Other; p = 0.9403, Mixed Models Repeated Measures; Mean Difference (Net) = 0.07, 95% CI 2-sided [-1.71 to 1.85]
Statistical Analysis 6: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 4; Test type: Superiority or Other; p = 0.5206, Mixed Models Repeated Measures; Mean Difference (Net) = -0.58, 95% CI 2-sided [-2.36 to 1.20]
Statistical Analysis 7: Comparison: Placebo vs Orvepitant 30 mg; Placebo Vs Orvepitant 30 mg at Week 6; Test type: Superiority or Other; p = 0.7140, Mixed Models Repeated Measures; Mean Difference (Net) = -0.36, 95% CI 2-sided [-2.30 to 1.58]
Statistical Analysis 8: Comparison: Placebo vs Orvepitant 60 mg; Placebo Vs Orvepitant 60 mg at Week 6; Test type: Superiority or Other; p = 0.0234, Mixed Models Repeated Measures; Mean Difference (Net) = -2.26, 95% CI 2-sided [-4.22 to -0.31]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAE) and non-serious adverse events (nSAE) were collected from Screening (Visit1), at Baseline (Day 1, Visit 2) until follow-up (Day 28, Visit 5).
Description: SAEs and nSAE are reported for all subjects population which comprised of all participants who received at least one dose of study medication.
Arm/Group | Placebo | Orvepitant 30 mg | Orvepitant 60 mg
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/113 | 0/107
Serious Adverse Events (participants affected / at risk) | 1/108 | 0/113 | 1/107
Other Adverse Events (participants affected / at risk) | 27/108 | 40/113 | 34/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=108) | Orvepitant 30 mg (N=113) | Orvepitant 60 mg (N=107)
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=108) | Orvepitant 30 mg (N=113) | Orvepitant 60 mg (N=107)
Headache (Nervous system disorders) | 10 | 11 | 5
Somnolence (Nervous system disorders) | 2 | 9 | 9
Dizziness (Nervous system disorders) | 3 | 7 | 2
Diarrhoea (Gastrointestinal disorders) | 7 | 9 | 7
Nausea (Gastrointestinal disorders) | 6 | 9 | 5
Dry mouth (Gastrointestinal disorders) | 6 | 8 | 4
Fatigue (General disorders) | 2 | 0 | 9
Upper respiratory tract infection (Infections and infestations) | 6 | 3 | 5

LIMITATIONS AND CAVEATS:
The study was terminated early upon recommendation of IDMC that was reviewing data from this trial and two other ongoing trials with same drug. When the trial was terminated 331 participants were randomized, compared to a target of 348 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.